CLINICAL TRIAL: NCT06716996
Title: Repeated Transcranial Magnetic Stimulation for the Treatment of Post-COVID Associated Affective Symptoms
Brief Title: RTMS for the Treatment of Post-COVID Associated Affective Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flurin Cathomas (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Flurin Cathomas, PD Dr. med., Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS-CO
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Post COVID -19 Depression
Keywords: Post COVID -19 depression; repeated transcranial magnetic stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS (Experimental)
  Interventions: Device: repeated transcranial magnetic stimulation
- sham treatment (Placebo Comparator)
  Interventions: Device: sham treatment

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation — 20 sessions of repeated transcranial magnetic stimulation
  Other Names: rTMS
  Arms: rTMS
Device: sham treatment — 20 sessions of sham treatment
  Arms: sham treatment

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) can lead to major post-acute sequelae. It is estimated that over 60 million people worldwide are affected by this multisystemic condition, here referred to as post-COVID. Affective symptoms such as fatigue and depressed mood are particularly prevalent in patients with post-COVID and pose significant individual and socioeconomic burdens. This stands in stark contrast to the currently limited number of available therapeutic options. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation modality that has been demonstrated to be both safe and effective in treating various neuropsychiatric disorders, including depression. However, whether rTMS also has an effect on post-COVID associated affective symptoms remains to be elucidated.

The overall objective of this randomized, double-blinded study is twofold: First, the investigators will examine the effect of rTMS on post-COVID associated affective symptoms. 52 individuals with post-COVID will be randomized to either receive 20 sessions of rTMS or sham treatment. A detailed psychopathological assessment of the study participants will be performed before and after the completion of rTMS/sham treatment. Secondly, the investigators will perform detailed characterization of the immune system before and after rTMS/sham treatment.

The individual burden and socioeconomic costs of post-COVID-associated neuropsychiatric symptoms are enormous, however, treatment options are limited. The investigators believe that the current proposal will address this key gap in the literature by testing whether rTMS, which constitutes a novel treatment with little side effects, could alleviate these debilitating symptoms. If proven effective, this study could pave the way for a completely new way in which post-COVID conditions are treated.

ELIGIBILITY:
Inclusion:

* Informed Consent as documented by signature
* Age between 18-65 years
* Proof of past COVID-19 infection by polymerase chain reaction (PCR) test or serology
* Negative COVID- 19 PCR test at the time of inclusion
* Affective symptoms (≥ 15 points on the Montgomery- Åsberg Depression Rating Scale) lasting for more than 12 weeks since COVID-19 infection
* No psychiatric history prior to the COVID-19 infection
* No major somatic comorbidities or substance use disorder

Exclusion:

* Contraindications to the rTMS treatment e.g. cochlear implants and metallic devices close to the TMS coil, a history of strokes, head injuries or seizures/epilepsy
* Epileptiform potentials in the electroencephalogram (EEG)
* Previous rTMS prior to the study
* Known severe hypersensitivity or severe adverse reaction to rTMS
* Women who are pregnant or breastfeeding
* Intention to become pregnant during the course of the study
* Psychiatric history prior to the COVID-19 infection
* Major somatic comorbidities e.g. renal failure, hepatic dysfunction, heart failure, cardiovascular disease.
* If the participant took antidepressants before the beginning of the study, there needs to be a washout period. The antidepressant has to be stopped for at least 3 weeks before commencing the study.
* The following drugs are not allowed during the study: any antidepressants, any antipsychotics, any drugs that lower the seizure threshold
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems
* Participation in another study with investigational treatment within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Depression severity | overall up to 13 weeks depending on the amount of rTMS/sham sessions per week (including a 4 week follow up)
  Depression severity will be assessed with the Montgomery-Åsberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Individual symptom dimensions and levels of functioning/quality of life. | overall up to 13 weeks depending on the amount of rTMS/sham sessions per week (including a 4 week follow up)
  Secondary outcomes will be clinical variables such as individual symptom dimensions and levels of functioning/quality of life.
Immune markers | overall up to 9 weeks depending on the amount of rTMS/sham sessions per week (biological variables will not be measured at the 4 week follow up)
  Blood-based biological variables of the immune system

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided